CLINICAL TRIAL: NCT04540562
Title: Evaluating the Feasibility of a Mobile Self-management Application for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Evaluating a Mobile Self-management Application for Patients With COPD Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-1257
Record Dates: First submitted 2020-08-25; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: mHealth; Self-management; Blended care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The COPD app consisted of an 8 week self-management program. The app had three views: timeline, information page, and contact page. The timeline was classified in 8 weeks, and each week included the lung exacerbation plan, daily and extra medication, information and education and questionnaires. The first week also included a video of a pulmonologist explaining the purpose of the app and additional information about the functionalities of the COPD app. A video consultation was planned after after 4 weeks and a face-to-face consultation after 8 weeks.
  Interventions: Other: COPD app

INTERVENTIONS:
Other: COPD app — The COPD app consisted of an 8 week self-management program. The app had three views: timeline, information page, and contact page. The timeline was classified in 8 weeks, and each week included the lung exacerbation plan, daily and extra medication, information and education and questionnaires. The first week also included a video of a pulmonologist explaining the purpose of the app and additional information about the functionalities of the COPD app. A video consultation was planned after after 4 weeks and a face-to-face consultation after 8 weeks.

SUMMARY:
The objective of the study is to evaluate the effects of a mobile self-management app in clinical practice for recently discharged COPD patients on application use, self-management, anxiety and depression, expectations and experiences, patients' and health care professionals' satisfaction and hospital readmissions.

DETAILED DESCRIPTION:
Usability testing techniques were used to receive feedback on a prototype of the app, before starting the feasibility study. Patients were recruited from a large teaching hospital. The COPD app provided patients with an 8 week self-management program. The application had three views: timeline, information page, and contact page. The start date was each patients' date of discharge. The timeline was classified in 8 weeks, and each week included the lung exacerbation plan, daily and extra medication, information and education and questionnaires. The first week also included a video of a pulmonologist explaining the purpose of the app and additional information about the functionalities of the COPD app. The timeline consisted of the lung exacerbation action plan, medication overview, weekly questionnaires and monitoring, and consultations (video consultation after 4 weeks and face-to-face consultation after 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Years
* Diagnosed with COPD
* Admissions to the hospital for exacerbation
* Having (access to) a tablet or smartphone
* Working internet connection
* Proficiency in using a tablet or smartphone
* Ability to read and understand the Dutch language
* Signed informed consent
* At least one hospitalization for COPD exacerbation in the year preceding the study (outcome was...)

Exclusion Criteria:

* No exacerbation of COPD
* Comorbidities: cancer, severe cognitive or psychiatric comorbidities
* No access to a tablet or smartpone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Use (feasibility) | Week 1 through week 20
  Use based on log data: number of times the app was used per week.
Satisfaction (feasibility) | Week 8
  Questionnaires were used to assess satisfaction, information and user-friendliness of the app. The items were rated on a 7 point scale, varying from 1 (totally disagree) to 7 (totally agree). Overall satisfaction was rated on a scale from 1 (very unsatisfied) to 10 (very satisfied). Multiple response questions were used to assess if patients missed information in the app. Suggestions for improvement were asked using an open question. Yes/no questions were used to assess satisfaction with video consultation(s) (additional requested video consultations, problems and time saving).
Overall satisfaction (feasibility) | Week 20
  Overall satisfaction was rated on a scale varying from 1 (not satisfied) to 10 (very satisfied). Suggestion for improvement were assessed with an open question.

SECONDARY OUTCOMES:
Self-management - change over time | Baseline, week 8 and week 20
  Self-management using Partner in Health Scale. The items are rated on a 9-point Likert scale varying from 0 (low self-management) to 8 (high self-management).
Expectations | Baseline
  Expectations with technology: using questions covering constructs of Unified Theory of Acceptance and Use of Technology. The items were rated on a 7 point scale varying from 1 (totally disagree) to 7 (totally agree).
Experiences with technology | Week 8
  Experiences with technology: using questions covering constructs of Unified Theory of Acceptance and Use of Technology. The items were rated on a 7 point scale varying from 1 (totally disagree) to 7 (totally agree).
Experiences with technology | Week 20
  Experiences with technology: using questions covering constructs of Unified Theory of Acceptance and Use of Technology. The items were rated on a 7 point scale varying from 1 (totally disagree) to 7 (totally agree).
Anxiety - change over time | Week 1 until week 8
  Hospital Anxiety and Depression Scale. Seven items were rated on a 4 points Likert scale, varying from 0 (lowest anxiety level) to 3 (highest anxiety level).
Depression - change over time | Week 1 and Week 8
  Hospital Anxiety and Depression Scale. Seven items were rated on a 4 points Likert scale, varying from 0 (lowest depression level) to 3 (highest depression level).
Satisfaction nurses | After intervention completion, up to 15 months.
  Questions to assess nurses' experiences with the application, satisfaction, time investment and integration in their work process. The items were rated on a 5 point scale, varying from 1 (totally disagree) to 5 (totally agree). Overall satisfaction was rated on a scale from 1 (not satisfied) to 10 (very satisfied).
Hospital readmissions | 30 days
  Hospital admissions for at least 24 hours. The number of hospital admissions was obtained from the Electronic Medical Record. This was compared with the readmission rate from the previous year, November 2017 until November 2018.
Hospital readmissions | 8 weeks
  Hospital admissions for at least 24 hours. The number of hospital admissions was obtained from the Electronic Medical Record. This was compared with the readmission rate from the previous year, November 2017 until November 2018.
Hospital readmissions | 20 weeks
  Hospital admissions for at least 24 hours. The number of hospital admissions was obtained from the Electronic Medical Record. This was compared with the readmission rate from the previous year, November 2017 until November 2018.
Use | Week 8
  Questions about use of the application: number of times and time in minutes (multiple choice question), use of the different functionalities and which functionality is most important (multiple response question), if patients experienced problems (yes/no), received help using the application (yes/no) and if people in their environment helped them using the app (yes/no).
Use | Week 20
  Questions about use of the application: number of times and time in minutes (multiple choice question), use of the different information items and which item is most important (multiple response question), if patients experienced problems (yes/no), received help using the application (yes/no) and if people in their environment helped them using the app (yes/no).

OTHER OUTCOMES:
Age | Baseline
  Age extracted from Electronic Medical Record.
Education | Baseline
  Multiple choice question.
Partner | Baseline
  Living together with a partner (yes/no question).
Children | Baseline
  Having children (yes/no question).
Internet use (duration) | Baseline
  Multiple choice question, varying from less than six months to more than 3 years
Frequency internet use | Baseline
  Multiple choice question, varying from every day to never.
Tablet/smartphone skills | Baseline
  Question with 5 point scale varying from 1 (very bad) to 5 (very good).
Help needed to use app on smartphone/tablet | Baseline
  Yes/no question. If yes: open question to answer who was asked for help.

CONTACTS AND LOCATIONS:
Overall Officials: Wim van Harten, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kooij L, Vos PJE, Dijkstra A, van Harten WH. Effectiveness of a Mobile Health and Self-Management App for High-Risk Patients With Chronic Obstructive Pulmonary Disease in Daily Clinical Practice: Mixed Methods Evaluation Study. JMIR Mhealth Uhealth. 2021 Feb 4;9(2):e21977. doi: 10.2196/21977. PMID 33538699

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT04540562/Prot_SAP_000.pdf